CLINICAL TRIAL: NCT06432738
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose-escalation Design to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and QTc Effect Research
Brief Title: ZL-82 Double-blind Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL82-H-Ib
Record Dates: First submitted 2024-03-24; First posted 2024-05-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 600mg ZL-82 (Experimental): The subjects in the single-dose group were fasted and water-free for at least 10 hours the night before the administration. On the first day of the study (D1), the subjects were given ZL-82 tablets or placebo according to the requirements of the random table, and were followed as per the study. Schedule safety inspections and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; complete a series of safety inspections, PK, and PD sample collection on the 3rd day and leave the clinical trial facility on the 7th day Safety follow-up.
  Interventions: Drug: ZL-82
- 600mg ZL-82 placebo (Placebo Comparator): The subjects in the single-dose group were fasted and water-free for at least 10 hours the night before the administration. On the first day of the study (D1), the subjects were given ZL-82 tablets or placebo according to the requirements of the random table, and were followed as per the study. Schedule safety inspections and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; complete a series of safety inspections, PK, and PD sample collection on the 3rd day and leave the clinical trial facility on the 7th day Safety follow-up.
  Interventions: Drug: ZL-82 placebo
- 50mg ZL-82 (Experimental): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82
- 50mg ZL-82 placebo (Placebo Comparator): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82 placebo
- 100mg ZL-82 (Experimental): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82
- 100mg ZL-82 placebo (Placebo Comparator): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82 placebo
- 200mg ZL-82 (Experimental): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82
- 200mg ZL-82 placebo (Placebo Comparator): Subjects in the multiple-dose group were fasted and water-free for at least 10 hours the night before dosing, and were given ZL once a day according to the random table requirements from day 1 (D1) to day 10 (D10) of the study. -82 tablets or placebo, and undergo safety inspections according to the study schedule and complete PK, PD, and Holter collection according to the PK, PD, and Holter collection schedule; after completing a series of safety inspections, PK, and PD sample collection on day 12 Safety follow-up was conducted on day 16 after leaving the clinical trial facility.
  Interventions: Drug: ZL-82 placebo

INTERVENTIONS:
Drug: ZL-82 — This group of subjects take ZL-82
  Other Names: 600mg ZL-82; 50mg ZL-82; 100mg ZL-82; 200mg ZL-82
  Arms: 100mg ZL-82; 200mg ZL-82; 50mg ZL-82; 600mg ZL-82
Drug: ZL-82 placebo — This group of subjects take ZL-82 placebo
  Other Names: 600mg ZL-82 placebo; 50mg ZL-82 placebo; 100mg ZL-82 placebo; 200mg ZL-82 placebo
  Arms: 100mg ZL-82 placebo; 200mg ZL-82 placebo; 50mg ZL-82 placebo; 600mg ZL-82 placebo

SUMMARY:
ZL-82 tablets are highly selective covalent irreversible inhibitors of non-receptor tyrosine protein kinase 3 (Janus kinase 3, JAK3) developed by Chengdu Zenitar Biomedical Technology Co., Ltd. According to Document No. 44 of 2020 "Chemical Drug Registration Classification and Application Document Requirements", it belongs to Category 1 chemical drugs and is an innovative drug that has not been marketed at home or abroad.

ZL-82 tablets have completed non-clinical pharmacology, non-clinical PK, and toxicology experiments, and have obtained the first-in-human randomized double-blind, placebo-controlled, dose-increasing dose-increasing approval for single oral administration of ZL-82 tablets. Partial results of the phase I clinical study on safety tolerability, pharmacokinetics and preliminary pharmacodynamics. It is necessary to further explore the safety, tolerability, pharmacokinetics and pharmacodynamic characteristics of multiple administrations based on the results obtained from the first human trial.

Non-clinical in vitro hERG tests and in vivo animal safety pharmacology tests of ZL-82 tablets showed no relevant cardiac safety concerns. According to the ICH E14 guideline "Clinical Evaluation of QT/QTc Interval Prolongation and Potential Proarrhythmic Effects of Non-Antiarrhythmic Drugs" Evaluation》2, it is recommended to conduct cardiac safety evaluation of experimental drugs with systemic bioavailability to evaluate the impact of experimental drugs on cardiac safety. This evaluation should include evaluation of the effect of the new drug on the QT/QTc interval and collection of adverse cardiovascular events. Establishing a relationship between ZL-82 drug concentration and QT/QTc interval changes will provide additional information for the analysis of cardiac repolarization trial planning and interpretation to facilitate analysis of the effects of drugs on QT/QTc interval changes. Concentration-response analysis, used to characterize the effect of the test drug on the QT/QTc interval, can be used as an alternative to time point analysis.

This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic characteristics of ZL-82 tablets in single/multiple oral doses in healthy subjects, and will also evaluate the effect of ZL-82 tablets on QTc.

ELIGIBILITY:
Inclusion Criteria:

1. Those who can understand the informed consent form, voluntarily participate in the trial and sign the informed consent form.
2. Male or female; aged between 18 and 50 years old (including 18 and 50 years old).
3. Male subjects weigh >=50kg, female subjects weigh >=45kg, body mass index (BMI) between 19.0~26.0kg/m^2, BMI = weight (kg)/height^ 2 (m^2), including boundary values.
4. The subject can communicate well with the researcher and complete the trial in compliance with the requirements of the protocol.

Exclusion Criteria:

-

Subjects who meet any of the following criteria will be excluded from the trial:

Current medical history, past medical history, and recent medication history:

1. Those who have a history of severe systemic diseases (including cardiovascular system, digestive system, urinary system, respiratory system, etc.), mental illness, and drug dependence;
2. Have a history of structural heart disease, heart failure, myocardial infarction, angina pectoris, torsade de pointes, ventricular tachycardia, QT prolongation syndrome or symptoms of QT prolongation syndrome (such as syncope) , convulsions) and family history (proven hereditary or close relatives died suddenly due to cardiac causes when young);
3. Physical examination, vital signs, laboratory examination items and test-related examinations and tests during the screening period or baseline period (for example: chest X-ray examination, abdominal color ultrasound, blood pregnancy test, ANA examination, gamma-interferon release Test, 12-lead electrocardiogram, etc.) with abnormal results and clinical significance;
4. Patients with a history of lipid metabolism defects, such as: familial hyperlipidemia, lipoid nephropathy, or patients with acute pancreatitis accompanied by hyperlipidemia;
5. Nervous/psychiatric, respiratory system, cardiovascular system, digestive tract system, blood and lymphatic system, endocrine system, musculoskeletal system diseases, liver and kidney dysfunction, or any other diseases and physiological conditions that may affect the test results during screening By;
6. Those with allergies, or those with a history of food or drug allergies or other allergic diseases (asthma, urticaria, eczematous dermatitis, etc.) that are clinically significant as determined by the researcher; or those who are known to be allergic to JAK inhibitors or to the test Those who are allergic to the excipients contained in the medicine;
7. Those who have suffered from clinically significant diseases or undergone major surgeries within 3 months before screening;
8. Those who suffered from acute diseases within 2 weeks before screening; those who had clinically significant infections within 3 months before screening (such as upper respiratory tract infection, nasopharyngitis, urinary tract infection, etc.); those who had any evidence of infection within 7 days before screening (such as Fever, cough, sputum, headache, etc.); those with a history of herpes simplex infection or recurrent (>1 time) herpes zoster or disseminated herpes zoster;
9. Those with a history of dysphagia or any gastrointestinal system disease (or gastrointestinal resection, etc.) that affects drug absorption;
10. Those who have donated blood within 3 months before screening, or those who plan to donate blood during this trial, or those who have had blood transfusion or blood loss ≥ 200mL within 4 weeks before the trial;
11. Those who have participated in 4 or more clinical trials as subjects in the past year; or those who have participated in any clinical trials as subjects within 3 months before participating in this trial;
12. Those who have a history of drug abuse within 5 years before screening or have used drugs within 3 months before screening;
13. Concomitant use of strong inducers of liver metabolic enzymes (such as: omeprazole, barbiturates, carbamazepine, aminoglutethimide, griseofulvin, promethazine) within 4 weeks (28 days) before screening esters, phenytoin, gramide, rifampicin, sulfinpyrazone, roxithromycin, etc.); those who have taken any drug known to cause QT/QTc interval prolongation within 4 weeks (28 days) before screening or have Medications that pose a risk of torsade de pointes (TdP);
14. Those who have been vaccinated within 8 weeks before screening, or plan to be vaccinated during the study or within 8 weeks after the last dose of study drug;
15. Those who have a history of fainting from blood and needles and cannot tolerate blood collection with intravenous indwelling needles;

    Health status:
16. Those whose 12-lead electrocardiogram during the screening period or baseline period has the following results: QTcF interval corrected according to Fridericia's formula >450ms; or those whose electrocardiogram is abnormal and the researcher believes that the abnormality is clinically significant (including but not limited to complete left bundle branch or right bundle branch block; second or third degree atrioventricular block (AVB); sustained atrial or ventricular arrhythmias; two consecutive ventricular premature contractions; ST-segment elevation pattern and myocardial ischemia Consistent; evidence of previous myocardial infarction (MI), left ventricular hypertrophy (LVH), or more than mild nonspecific ST-T wave changes; any features that make QT assessment unreliable, including flattened T waves);
17. Those with systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg during the screening period or baseline period;
18. Laboratory test results during the screening period or baseline period that the researcher considers to be abnormal and clinically significant, including but not limited to:

    1. Abnormal renal function during the screening period or baseline period: serum creatinine > upper limit of normal (ULN) or glomerular filtration rate (GFR, calculated by CKD-EPI formula) <90mL/min/1.73m2;
    2. Direct bilirubin and total bilirubin>1.5xULN;
19. Those who are positive for hepatitis B virus surface antigen and/or positive for hepatitis B virus e antigen, positive for hepatitis C virus antibodies, positive for human immunodeficiency virus antibodies, or have abnormal Treponema pallidum antibodies during the screening period;
20. Those who have a positive alcohol breath test during the screening period or baseline period, or a positive urine drug abuse screen;

    Lifestyle restrictions:
21. Have special requirements for diet and cannot comply with the diet and corresponding regulations provided by clinical research institutions;
22. Those who cannot control special diets (including dragon fruit, mango, grapefruit and/or xanthine diets, caffeinated foods or beverages, etc.) from 48 hours before the first dose to the end of the study;
23. Those who have taken special diets or exercised strenuously within 48 hours before the first dose, or have other factors that affect drug absorption, distribution, metabolism, excretion, etc.;
24. Regular drinkers within 6 months before administration or during the trial, that is, drinking more than 21 units (men) or 14 units (women) of alcohol per week (1 unit = 360mL beer or 45mL liquor with an alcohol content of 40%) or 150mL wine);
25. Those who smoked more than 5 cigarettes per day in the 3 months before administration, or who will use any tobacco products during the trial; contraception:
26. Pregnant or lactating women or those with positive blood pregnancy test results;
27. Those who have used long-acting estrogen or progesterone injections or implants within 6 months before screening;
28. Women of childbearing age who had unprotected sex with their partners within 14 days before screening;
29. Male or female subjects of childbearing potential do not agree to use effective contraceptive methods from the time of signing the informed consent form to 6 months after the last dose.

    Other standards:
30. Subjects who the researcher believes have poor compliance or have any factors that are not suitable for participating in this trial;
31. Relevant personnel of the research center and their family members;
32. Vulnerable subjects such as students and subordinates of researchers and employees of sponsors;
33. Subjects may not be able to complete this trial due to other reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
ZL-82 Pharmacokinetics (PK)：Cmax | 72hours
  security indicators
ZL-82 Pharmacokinetics (PK)：Tmax | 72hours
  Estimation of time to reach Cmax
ZL-82 Pharmacokinetics (PK)：AUC0-72h | 72hours
  Estimation of AUC from time zero to the last measured time point
ZL-82Pharmacokinetics (PK)：AUC0-∞ | 72hours
  Estimation of AUC from time zero extrapolated to infinity
ZL-82 Pharmacokinetics (PK)：MRT | 72hours
  Estimation of mean residence time
ZL-82 Pharmacokinetics (PK)：Vd | 72hours
  Estimation of apparent volume of distribution
ZL-82 Pharmacokinetics (PK)：t1/2 | 72hours
  Estimation of terminal elimination half-life
ZL-82 Pharmacokinetics (PK)：CLz/F | 72hours
  Estimation of clearance when dosed orally

SECONDARY OUTCOMES:
Evaluation of the pharmacodynamic (PD) characteristics of single/multiple oral doses of ZL-82 tablets in healthy humans | Day 16
  security indicators
To evaluate the effect of ZL-82 tablets on QT/QTc interval in healthy subjects after single-dose administration. | Day 16
  security indicators
To evaluate the effect of ZL-82 tablets on ECG parameters (ΔQTcF/ΔΔQTcF and HR, PR, QRS intervals) in healthy subjects, as well as the effect on T wave morphology and U wave. | Day 16
  security indicators

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Medical Shandong Hospital of Traditional Chinese Medicine, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No